CLINICAL TRIAL: NCT05145972
Title: Efficacy of Adding Lidocaine 10% to Phenol in Ultrasound Guided Superior Hypogastric Plexus Neurolysis in The Management of Pelvic Cancer Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, assist. prof. of anesthesia and pain management, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MS.21.04.1458
Record Dates: First submitted 2021-11-12; First posted 2021-12-06 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Efficacy of Adding Lidocaine 10% to Phenol in Superior Hypogastric Plexus Neurolysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- • Group P (Active Comparator): Ultrasound guided SHPN will be done by injecting 10 ml of Phenol 10 %.
  Interventions: Other: Ultrasound Guided Superior Hypogastric Plexus
- • Group LP (Active Comparator): Ultrasound guided SHPN will be done by injecting 10 ml Phenol 10 % then injecting 3 ml Lidocaine 10%.
  Interventions: Other: Ultrasound Guided Superior Hypogastric Plexus

INTERVENTIONS:
Other: Ultrasound Guided Superior Hypogastric Plexus — The division of abdominal aorta into common iliac arteries will be identified by using longitudinal sonography , and the body of the fifth (5th) Lumbar vertebra will be identified by placing the transducer transversely. A skin wheal will be raised with subcutaneous infiltration with 2% lidocaine solution nearly 3-4 cm below the umbilicus. A 15-cm Long 22-G Chiba needle will be used with out of plane technique, and the needle will be advanced under USG-guidance to reach the anterior- most point of the fifth Lumber vertebral body avoiding the vascular structures. The needle will be withdrawn nearly 1-2 mm after hitting the vertebral body to avoid injecting the drug into the periosteum. After confirming a negative aspiration of blood, known amount of neurolytic agent according to the grouping will be injected for the neurolysis of superior hypogastric plexus. The uniform spread of the drug will be confirmed under real-time sonography.

SUMMARY:
The superior hypogastric plexus (SHP) is a complex nervous collection located at the lumbosacral region below the level of the aortic bifurcation at the level of the lower third of the fifth lumbar vertebral body and upper third of the first sacral vertebral body at the sacral promontory Neurolytic agents, such as alcohol and phenol have been used to ablate peripheral nerves to treat pain and spasticity . These agents were nonspecific for neuronal tissue and complications have been seen involving damage to surrounding soft tissue (skin, muscle, vascular) and pain on alcohol injection

Lidocaine has been demonstrated to be neurotoxic in high concentrations at 10% and can be used as a neurolytic agent with no effect on motor function, muscle state, or surrounding tissue rather than other neurolytic.

DETAILED DESCRIPTION:
Every Patient will be in supine Trendelenburg position, IV access in case of adverse events and for moderate sedation if needed (for patient comfort, sever anxiety or needle phobia, or history of vagal events).

The procedure will be completed under aseptic precautions. The division of abdominal aorta into common iliac arteries will be identified by using longitudinal sonography (Lumify L12-4 Linear Array Transducer 12 to 4 MHz extended operating frequency range, 34mm footprint and aperture size, and scan depth of up to 12cm. Imaging modes include 2D, color Doppler, and M-mode), and the body of the fifth (5th) Lumbar vertebra will be identified by placing the transducer transversely. A skin wheal will be raised with subcutaneous infiltration with 2% lidocaine solution nearly 3-4 cm below the umbilicus. A 15-cm Long 22-G Chiba needle will be used with out of plane technique, and the needle will be advanced under USG-guidance to reach the anterior- most point of the fifth Lumber vertebral body avoiding the vascular structures. The needle will be withdrawn nearly 1-2 mm after hitting the vertebral body to avoid injecting the drug into the periosteum. After confirming a negative aspiration of blood, known amount of neurolytic agent according to the grouping will be injected for the neurolysis of superior hypogastric plexus. The uniform spread of the drug will be confirmed under real-time sonography. Vital Sign parameters will be recorded during and after the procedure, during which patients remained fully awake

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years old.
* Either genders.
* Cancer-related pelvic pain.
* American Society of Anesthesiologists Physical Status class I and II.
* Patients receiving opioids for pelvic cancer pain with visual analogue pain scale more than 4.
* BMI < 30.

Exclusion Criteria:

* . patient refusal. local or systemic sepsis. Coagulopathy. unstable cardiovascular and respiratory diseases. previous neurological deficits, history of psychiatric disorders history of drug abuse distorted local anatomy. allergy to the used medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-30 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
: NRS | after 1 week from block
  from 0 to 10 (0= no pain ,10 =maximum pain)
NRS | after 1 month from block
  from 0 to 10 (0= no pain ,10 =maximum pain)
NRS | after 2 month from block
  from 0 to 10 (0= no pain ,10 =maximum pain)
NRS | after 3 month from block
  from 0 to 10 (0= no pain ,10 =maximum pain)

SECONDARY OUTCOMES:
Patient satisfaction | after injection
  using a linear scale in which 0 is unsatisfied and 1
daily analgesic requirements | after 3 months from injection
  the patient need of analgesia tramandin 100mg after injection
side effect during injection | during injection
  any complication during injection as hemorrhage and hypotension